CLINICAL TRIAL: NCT04132310
Title: Pregnancy Weight Trajectories and Offspring Adiposity
Brief Title: Mother Infant Nutrition Study
Acronym: MINT
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Elizabeth Widen, Assistant Professor, University of Texas at Austin
Other Study IDs: R00HD086304 (NIH)
Record Dates: First submitted 2019-10-10; First posted 2019-10-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Related; Infant Development
Keywords: Pregnancy; body composition; infant adiposity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal biospecimen samples collected: blood (serum and plasma), urine, microbiome, breastmilk, placenta, umbilical cord and cord blood.
  Infant biospecimen samples collected: saliva, meconium, transitional stool, fecal sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MINT Participants: Up to 60 MINT maternal participant are linked with 60 infant participants, and 60 partner participants.
  Interventions: Other: N/A This is an observational study.

INTERVENTIONS:
Other: N/A This is an observational study. — This is an observational study.

SUMMARY:
Early life influences (including the intrauterine environment, birth weight, and early postnatal growth) shape subsequent weight trajectories and future chronic disease risk. The MINT study will evaluate whether maternal fat mass changes are associated with specific maternal weight trajectories during pregnancy, and with neonatal adiposity at birth. The study is a prospective observational cohort currently enrolling women in early pregnancy,and following mothers and infants after birth.

DETAILED DESCRIPTION:
The Institute of Medicine (IOM) recommendations were established with limited evidence showing how the pattern of weight gain is associated with short-and long-term health of mothers and their children. Previous studies evaluated the impact of overall gestational weight gain pattern across gestation using latent class analysis and others have evaluated maternal weight change pattern-by trimester or early/late pregnancy-on offspring size and adiposity. However, it remains unclear if there are weight gain trajectories or specific periods of weight gain that are associated with greater adiposity in offspring, and whether effects persist across the life course.

The MINT study will expand our understanding of determinants that are influencing maternal weight trajectories, including race/ethnicity, prepregnancy BMI and parity. Although many factors are well-established determinants of pregnancy weight gain, such as prepregnancy BMI and parity, there is limited understanding of whether these factors and others, such as maternal diet, race, psychosocial health or socio-economic status, influence the overall pattern of pregnancy weight gain and the IOM has called for research in this area. This knowledge is essential for providing personalized clinical recommendations for weight gain monitoring and to develop interventions to support healthy weight gain that optimizes health outcomes for mother and child.

This study is an observational, prospective cohort design, and will recruit up to 60 volunteers with singleton gestations of BMI 18.5-35. The mothers' will be assessed at 14-15, 24-25, and 35 weeks of pregnancy, and at 6 weeks post-delivery. Additional measurements may also be collected at 6-, 12-, and 24-months postpartum. The measurements will include anthropometry (weight, height, circumferences, and skin fold thicknesses), and whole body magnetic resonance imaging (MRI) and/or dual-energy X-ray absorptiometry (DXA). The infants' measurements will be anthropometry at birth (2-3 days), and approximately 1 and 6 weeks. Additional measurements may also be collected at 6-, 12-, and 24-months. Infants will also undergo air displacement plethysmography (PeaPod) at approximately 1 week and 6 weeks, and potentially DXA at 12- and 24-months. Biospecimen samples will be collected, including: maternal serum, plasma, urine, microbiome, breastmilk, placenta, umbilical cord and cord blood, infant meconium and stool, and infant saliva. Data will be collected regarding mothers' dietary intake and physical activity (questionnaires and accelerometry). Other data to be collected include questionnaires on quality of life, socio-economic status, health behaviors and intentions. If the woman identifies a partner, the partner will be invited to complete questionnaires on health, health behaviors and anthropometry measures.

ELIGIBILITY:
Inclusion Criteria:

1. <16 weeks gestation
2. Age >18 years old
3. BMI <35 kg/m2
4. Width <48 cm

Exclusion Criteria:

1. Diabetes
2. Claustrophobia
3. Recent weight loss of >5% of body weight before pregnancy
4. Weight-loss related surgery
5. Currently breastfeeding
6. Smoking
7. Presence of any mechanically or magnetically activated implants, or any other contraindication for MRI

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We plan to recruit up to 60 pregnant women around 8-14 weeks gestation and will follow the 60 babies after birth. If the pregnant mother identifies a partner for the partner component, we will seek to enroll the partner in the study, and therefore, we estimate that we will enroll up to 60 partners.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal fat mass changes during pregnancy and postpartum | 14, 24, 35 weeks gestation, and up to 24-months postpartum
  Mother's fat mass at 14 weeks, 24 weeks, and 35 weeks gestation, and up to 24-months postpartum as a continuous variable. This will be ascertained through MRI and DXA.
Infant percent fat at birth | 24-72 hours after birth
  Infant percent fat at birth as a continuous variable. This will be ascertained through neonatal skinfolds and anthropometry.

SECONDARY OUTCOMES:
Maternal weight trajectories during pregnancy and postpartum | Weekly after enrollment (up to 6 weeks postpartum), biweekly 2 to 24 months postpartum
  Mother's weekly weights will be modeled using trajectory modeling as a continuous variable.
Maternal regional adipose tissue during pregnancy and postpartum | 14, 24,35 weeks gestation, and up to 24-months postpartum
  Mother's weight at 14 weeks, 24 weeks, and 35 weeks gestation, and up to 24-months postpartum, as a continuous variable. This will be ascertained through anthropometry, DXA, and MRI.
Infant percent fat after birth | 1-week to 24-months
  Infant percent fat at 1-week, 6-weeks, 6-months, 12-months, and 24-months old as a continuous variable. This will be ascertained through anthropometry, PeaPod, and DXA.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Health Discovery Building Biomedical Imaging Center, Austin, Texas
  - Dell Pediatric Research Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Data will only be shared with individuals who are collaborating with the research team on this study; these investigators will be added to the IRB or only provided with a limited deidentified dataset. The data will not be destroyed.